CLINICAL TRIAL: NCT07291908
Title: Correlation of Inflammation Severity With Pulmonary Gas Exchange and MiRNA 126 in Trauma Patients
Brief Title: Inflammation Severity and miRNA-126 in Trauma
Status: Recruiting | Type: Observational
Sponsor: Melike Cengiz (Other)
Responsible Party: Sponsor-Investigator, Melike Cengiz, Prof Dr, Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: TBAEK-307
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Trauma ICU Patients; Endothelial Injury
Keywords: ARDS; MULTITRAUMA; MICRORNAS; ENDOTHEL

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with ARDS and Were Followed in ICU After Trauma: Patients who developed ARDS and were followed in intensive care for at least 3 days after trauma
- Patients without ARDS and Were Followed in ICU After Trauma: Patients who does not developed ARDS and were followed in intensive care for at least 3 days after trauma
- Control Group: Control group of healthy volunteers of similar age and gender

SUMMARY:
Trauma triggers a complex immune response intended to eliminate danger signals and restore physiological balance. Early post-traumatic inflammation is primarily initiated by damage-associated molecular patterns (DAMPs) and pathogen-associated molecular patterns (PAMPs). In patients with severe trauma, dysregulated inflammation increases susceptibility to infection, systemic inflammatory response syndrome (SIRS), multiple organ dysfunction syndrome (MODS), and mortality. The lungs are particularly vulnerable, and excessive inflammatory activation may lead to acute lung injury (ALI) or acute respiratory distress syndrome (ARDS), conditions characterized by increased vascular permeability, alveolar epithelial injury, surfactant dysfunction, and impaired gas exchange.

Pro-inflammatory cytokines, activated neutrophils, reactive oxygen species, and proteases contribute to endothelial and epithelial barrier disruption. Recent evidence also suggests that several microRNAs, including miR-126, may play a regulatory role in pulmonary barrier integrity through modulation of tight-junction proteins and PI3K/AKT-related pathways.

Although many components of the trauma-related inflammatory response have been described, the relationship between systemic inflammatory severity and impairment of pulmonary gas exchange remains insufficiently defined in clinical settings.

This study aims to investigate the correlation between inflammatory severity markers (C-reactive protein, procalcitonin, IL-6, reactive oxygen derivatives, neutrophil-to-lymphocyte ratio, lactate), imaging findings (flow-mediated dilation by ultrasound), clinical parameters (blood pressure, heart rate, urine output, vasoactive medication requirements), pulmonary gas-exchange measurements (arterial blood gases, PaO₂/FiO₂ ratio), and circulating miRNA-126 levels in trauma patients. The findings may help identify biomarkers that better reflect inflammatory burden and the risk of lung dysfunction following trauma.

DETAILED DESCRIPTION:
Trauma elicits a complex immune response aimed at eliminating perceived threats and restoring physiological homeostasis. This response is initiated through the activation of damage-associated molecular patterns (DAMPs) and pathogen-associated molecular patterns (PAMPs), which function as the initial "signal 0" in the inflammatory cascade. In trauma patients, the balance between pro-inflammatory and anti-inflammatory mediators may become dysregulated, resulting in heightened vulnerability to severe infections even from low-virulence microorganisms. Such dysregulation contributes to increased rates of systemic inflammatory response syndrome (SIRS), multiple organ dysfunction syndrome (MODS), and mortality. Elevated cytokine release and activation of macrophages and lymphocytes further intensify the inflammatory process and the severity of SIRS.

The lungs are particularly susceptible to inflammatory injury following trauma. Acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) represent major complications, characterized by increased vascular permeability and persistent pulmonary inflammation. Severe trauma, high thoracic injury scores, hypotension, metabolic acidosis, major fractures, and delays in treatment are factors known to contribute to ARDS development.

Under normal conditions, the lung maintains minimal alveolar fluid through a balance of vascular oncotic pressure, intact tight junctions, and effective lymphatic drainage. When this barrier is disrupted by trauma or inflammation, plasma proteins and fluid leak into the interstitium and alveolar spaces, leading to protein-rich pulmonary edema. Type I alveolar epithelial cells (AEC-I), which cover most of the alveolar surface and form a tight barrier essential for gas exchange, become damaged. Type II alveolar epithelial cells (AEC-II), responsible for surfactant production and epithelial repair, may lose function, resulting in alveolar collapse due to surfactant depletion. Consequently, lung compliance decreases, pulmonary arterial pressures rise, and ventilation-perfusion mismatch leads to hypoxemia.

The pathogenesis of ARDS involves multiple biological processes, including inflammation, apoptosis, and thrombosis. Early in the syndrome, pro-inflammatory cytokines such as TNF-α, IL-1, IL-6, and IL-8 are released. Neutrophils accumulate within the pulmonary microvasculature and alveolar spaces, where they release reactive oxygen species, proteases, and other cytotoxic mediators, causing further epithelial and endothelial injury.

In recent years, microRNAs (miRNAs) have emerged as potential regulators in ARDS and other inflammatory lung injuries. miR-126, in particular, has been found to be elevated in animal models of lipopolysaccharide-induced lung injury and within exosomes derived from human endothelial progenitor cells. Experimental studies suggest that miR-126 supports the integrity of alveolar and endothelial barriers by enhancing tight-junction protein expression (such as claudins and occludin) and modulating signaling pathways involving PIK3R2, HMGB1, VEGFα105, Rac1, and AKT. These findings indicate that miR-126 may have a protective role in maintaining pulmonary barrier function, although no miRNA-targeted therapy is currently approved for ARDS.

Despite the extensive understanding of trauma-induced inflammation, there is a lack of clinical research examining how the severity of systemic inflammation correlates with pulmonary gas-exchange impairment. Biomarkers such as C-reactive protein, procalcitonin, IL-6, reactive oxygen derivatives, and neutrophil-to-lymphocyte ratio, as well as clinical parameters including blood pressure, heart rate, urine output, and vasoactive medication requirements, are widely used to assess inflammatory status and physiologic stability. Imaging tools, such as flow-mediated dilation (FMD) measured by ultrasound, provide additional insight into endothelial function. However, their relationship with pulmonary gas-exchange indices-particularly arterial blood gases and the PaO₂/FiO₂ ratio-remains unclear.

This study is designed to investigate the correlations among laboratory markers of inflammation, bedside clinical measurements, endothelial imaging parameters, pulmonary gas-exchange data, and circulating miR-126 levels in trauma patients. By examining these relationships, researchers aim to identify biomarkers that may better reflect the severity of inflammation and the risk of lung dysfunction following trauma. Such insights may ultimately support more accurate prognostication and improved clinical management strategies for trauma-related pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older.

Patients monitored and treated for trauma in the anesthesia intensive care units of Akdeniz University Faculty of Medicine.

Exclusion Criteria:

Patients younger than 18 years.

Patients with concomitant thoracic trauma.

Presence of active infection prior to trauma.

Patients not admitted to the ICU within the first 24 hours after trauma.

Patients who remain in the ICU for less than 72 hours following trauma.

Current use of steroids, chemotherapy, or antibiotic therapy prior to ICU admission.

Patients with immunodeficiency.

Patients who are in shock prior to or during ICU admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) admitted to the anesthesia intensive care units of Akdeniz University Faculty of Medicine with blunt or penetrating trauma. The population represents early post-traumatic ICU admissions without thoracic injury, pre-existing infection, immunodeficiency, or other conditions that may alter the inflammatory response.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Serum miRNA-126 Levels and Severity of Lung Injury | First 3 days of ICU admission.
  Measurement of circulating miRNA-126 levels and their correlation with pulmonary gas-exchange impairment (PaO₂/FiO₂ ratio, arterial blood gas parameters).

SECONDARY OUTCOMES:
Serum IL-6 and Syndecan Levels | First 3 days of ICU admission.
  Daily blood sampling for measurement of IL-6 and Syndecan as markers of systemic inflammation and endothelial injury.
Flow-Mediated Dilation (FMD) by Ultrasound | Within first 3 days of ICU admission.
  Assessment of endothelial function by measuring brachial artery flow-mediated dilation.

CONTACTS AND LOCATIONS:
Overall Officials: Melike Cengiz, Prof Dr, Study Director — Department of Anesthesiology and Reanimation, Akdeniz University Hospital; Canberk Kurban, Resident Physician, Principal Investigator — Department of Anesthesiology and Reanimation, Akdeniz University Hospital; Şükran Burçak Yoldaş, Prof Dr, Principal Investigator — Department of Medical Biology, Akdeniz University Hospital; Ülkü Arslan, Specialist Physician, Principal Investigator — Department of Anesthesiology and Reanimation, Akdeniz University Hospital
Locations (1):
- Akdeniz University Hospital, Antalya, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) collected during the study, including clinical variables, laboratory results, hemodynamic measurements, imaging findings, biomarker data (including IL-6, Syndecan, and miRNA-126 levels), and gas-exchange parameters, will be made available for research purposes. No information that could directly identify participants will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Deidentified IPD and supporting documents will be available beginning 6 months after publication of the study results, and will remain accessible without a predefined end date.
Access Criteria: Data will be shared with qualified researchers upon reasonable request. Investigators requesting access must submit:
  A short research proposal outlining study aims
  Institutional affiliation
  Ethics committee approval (if applicable) Access will be granted following the execution of a Data Use Agreement (DUA) to ensure protection of patient confidentiality.

REFERENCES:
- [Result] Johansson PI, Henriksen HH, Stensballe J, Gybel-Brask M, Cardenas JC, Baer LA, Cotton BA, Holcomb JB, Wade CE, Ostrowski SR. Traumatic Endotheliopathy: A Prospective Observational Study of 424 Severely Injured Patients. Ann Surg. 2017 Mar;265(3):597-603. doi: 10.1097/SLA.0000000000001751. PMID 27144442
- [Result] Lee LK, Medzikovic L, Eghbali M, Eltzschig HK, Yuan X. The Role of MicroRNAs in Acute Respiratory Distress Syndrome and Sepsis, From Targets to Therapies: A Narrative Review. Anesth Analg. 2020 Nov;131(5):1471-1484. doi: 10.1213/ANE.0000000000005146. PMID 33079870